CLINICAL TRIAL: NCT03232502
Title: Pharmacogenetics in Primary Care Psychotropics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pending1
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Depression; Obsessive-Compulsive Disorder; Generalized Anxiety Disorder
MeSH Terms: conditions — Depression; Obsessive-Compulsive Disorder; Generalized Anxiety Disorder | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Diagnostic Test: Pharmacogenetic testing

INTERVENTIONS:
Diagnostic Test: Pharmacogenetic testing — Basic pharmacogenetic panel
  Arms: Intervention

SUMMARY:
Pragmatic trial of pharmacogenetic testing at the time of prescription for a selective serotonin reuptake inhibitor, tricyclic antidepressant or atypical antipsychotic. Does real time intervention improve patient outcomes?

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Prescribed a drug of interest for the first time

Exclusion Criteria:

* Previous pharmacogenetic testing available

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-08-15 (Estimated); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient oriented outcome1- Clinical Improvement | 6 months
  Clinically significant improvement as noted by physician (Subjective and PHQ-9)
Patient oriented outcome2- Adverse effects | 6 months
  Number of patients with specific, common side effects (from medical chart)
Patient oriented outcome3- Time to Improvement | Up to 6 months
  Days to clinical improvement (from medical chart)
Patient oriented outcome5- Visits | 6 months
  Total number of visits to clinic with medication titration required (from medical chart)

IPD SHARING:
Plan to Share IPD: Undecided